CLINICAL TRIAL: NCT04883138
Title: A Phase 1 Single Ascending Dose Study of a Recombinant Hyperimmune Polyclonal Antibody Against SARS CoV-2 (GIGA-2050) in Patients Hospitalized With COVID-19
Brief Title: Recombinant Hyperimmune Polyclonal Antibody (GIGA-2050) in COVID-19 Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped for commercial reasons.
Sponsor: GigaGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GG-GIGA-2050-001
Record Dates: First submitted 2021-05-04; First posted 2021-05-12 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: SARS CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — GIGA-2050

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, first in human (FIH) study utilizing a 3+3 design to assess the safety and pharmacology of single ascending doses (SAD) of GIGA-2050 in patients hospitalized with confirmed COVID-19.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 5 mg GIGA-2050 per kg BW (Experimental): Participants will receive a single IV infusion of 5 mg GIGA-2050 per kg BW
  Interventions: Drug: GIGA-2050
- 15 mg GIGA-2050 per kg BW (Experimental): Participants will receive a single IV infusion of 15 mg GIGA-2050 per kg BW, or as determined by SRC review
  Interventions: Drug: GIGA-2050
- 50 mg GIGA-2050 per kg BW (Experimental): Participants will receive a single IV infusion of 50 mg GIGA-2050 per kg BW, or as determined by SRC review
  Interventions: Drug: GIGA-2050

INTERVENTIONS:
Drug: GIGA-2050 — Recombinant Hyperimmune Polyclonal Antibody

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending IV dose administrations of GIGA-2050 in patients hospitalized with COVID-19.

DETAILED DESCRIPTION:
This is a Phase 1, first in human (FIH) study utilizing a 3+3 design to assess the safety and pharmacology of single ascending doses (SAD) of GIGA-2050 in patients hospitalized with confirmed COVID-19. Participants will receive a single intravenous (IV) infusion dose of GIGA-2050 and followed for safety, pharmacology and efficacy assessments during hospitalization, after discharge (if applicable), and through study discontinuation or end of study visit (Day 56).

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 18 years of age.
* Positive result of a SARS CoV-2 RNA diagnostic test result ≤48 hours before enrollment, warranting hospital admission as per Investigator's judgement.
* COVID-19 pneumonia findings on imaging (chest X-ray or CT Scan).
* Requires oxygen supplementation with FIO2 approximately 30% or greater administered by nasal cannula, mask, or NIV.
* Participants can be on other medication on-label to treat COVID-19 respiratory disease that the Investigator deems clinically relevant in combination with the study drug, including corticosteroids. Passage of 24 hours after administration of the EUA drug will be required prior to dosing GIGA-2050.
* Men or non-lactating female participants who are surgically sterile or post-menopausal, or a Woman of Childbearing Potential (WCBP) with a negative pregnancy test at screening willing to use highly effective contraception methods.

Exclusion Criteria:

* Acute respiratory failure requiring invasive mechanical ventilation or ECMO at enrollment.
* Systolic Blood Pressure (SBP) <110 mmHg or heart rate >120 bpm.
* Pre-existing heart failure or unstable angina or myocardial infarction in the last month prior to screening.
* Pre-existing chronic respiratory condition(s).
* Evidence of acute kidney injury, increase of serum creatinine of ≥1.5 x baseline, or urine output of <0.5mL/kg/hr sustained for at least 6 hours once volume repleted.
* Aspartate aminotransferase (AST) ≥2.5 x ULN, alanine aminotransferase (ALT) ≥2.5 x ULN, and/or total bilirubin >1.5 x ULN, or severe hepatic impairment.
* Known systemic hypersensitivity to recombinant antibody therapies.
* Female participant who is pregnant.
* Participant is expected to transfer to a non-investigative facility from the investigation site and cannot be monitored for compliance with protocol-required safety monitoring procedures.
* Participants who are currently participating or have participated in another clinical trial within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 up to Day 56
  Frequency of TEAEs graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence of dose limiting toxicities (DLTs) | Day 1 up to Day 3
  Frequency of DLTs at each dose level
Change from baseline of vital signs, physical examination, and clinical laboratory assessments | Day 1 up to Day 56
  Numeric summaries of all observed findings and changes for vital signs, laboratory assessments, physical examinations, and ECG
Incidence of infusion-related reactions (IRR) and hypersensitivity reactions | Day 1 through Day 2
  Frequency of IRR and hypersensitivity reactions

SECONDARY OUTCOMES:
Pharmacological evaluation of single doses of GIGA-2050 | Day 1 up to Day 28
  Serum titers of antibodies directed against SARS CoV-2 will be measured for the pharmacological profile of single doses of GIGA-2050

CONTACTS AND LOCATIONS:
Overall Officials: Sean Liu, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share IPD due to evaluation of potential DLTs.

REFERENCES:
- [Background] Keating SM, Mizrahi RA, Adams MS, Asensio MA, Benzie E, Carter KP, Chiang Y, Edgar RC, Gautam BK, Gras A, Leong J, Leong R, Lim YW, Manickam VA, Medina-Cucurella AV, Niedecken AR, Saini J, Simons JF, Spindler MJ, Stadtmiller K, Tinsley B, Wagner EK, Wayham N, Tracy L, Lundberg CV, Buscher D, Terencio JV, Roalfe L, Pearce E, Richardson H, Goldblatt D, Ramjag AT, Carrington CVF, Simmons G, Muench MO, Chamow SM, Monroe B, Olson C, Oguin TH, Lynch H, Jeanfreau R, Mosher RA, Walch MJ, Bartley CR, Ross CA, Meyer EH, Adler AS, Johnson DS. Generation of recombinant hyperimmune globulins from diverse B-cell repertoires. Nat Biotechnol. 2021 Aug;39(8):989-999. doi: 10.1038/s41587-021-00894-8. Epub 2021 Apr 15. PMID 33859400